CLINICAL TRIAL: NCT03118089
Title: Efficacy of a Nutrition Biscuit in Malnutrition Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/NI/1036
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Malnutrition
Keywords: Oral nutritional supplements
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biscuit style oral nutritional supplement treatment (Experimental): Participants will take the biscuit style oral nutritional supplement at an intervention level equivalent to their current oral nutritional supplement prescription
  Interventions: Dietary Supplement: Biscuit style oral nutritional supplement
- Standard Care (No Intervention): Participants will remain on their current oral nutritional supplement

INTERVENTIONS:
Dietary Supplement: Biscuit style oral nutritional supplement
  Arms: Biscuit style oral nutritional supplement treatment

SUMMARY:
The health risks and costs associated with malnutrition can be significantly reduced if symptoms are recognized early and treated effectively. Oral nutritional supplements (ONS) have been shown to increase nutrient intakes and maintain or improve nutritional status and functional outcomes in patients in a variety of settings. However despite this it is frequently reported that compliance to ONS, which are often milk based drinks, is poor. The aim of the present study is to assess the effectiveness of a new biscuit style nutritional supplement in the management of malnutrition.

The study is a randomized controlled eight-week intervention study. Suitable participants currently being prescribed ONS and who meet the study inclusion and exclusion criteria, will be identified by either staff in care facilities, Registered Dietitians or by General Practitioner (GP) surgeries. Participants (n=80) will be stratified based on BMI and gender and randomly assigned to either the biscuit ONS group (n=40) or to remain on their existing ONS prescribed as part of their standard care practice (n=40). Changes in anthropometry, functional status, nutritional intake and appetite, general health, gastrointestinal symptoms and biochemistry (correction of nutritional deficiency), as well as compliance and acceptability of ONS will be assessed between week 0 and week 8. Participants will also be visited mid-intervention (week 4) to ensure well-being and assess compliance.

This work is funded by Calerrific Ltd. and seeks to determine if the new biscuit style nutritional supplement could be used as an alternative to, or in conjunction with, existing ONS to improve compliance and aid the recovery of malnourished patients.

ELIGIBILITY:
Inclusion Criteria:

* Currently requiring oral nutritional supplement (minimum 8 weeks)

Exclusion Criteria:

* Requiring tube or parenteral nutrition, texture modification or specialised diet
* Diagnosed chronic renal or liver disease, diabetes T1, cancer cachexia
* Any other condition whereby taking part in the study may have a negative impact on well-being

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-10-30 (Estimated)

PRIMARY OUTCOMES:
Weight change | Change over 8 weeks from baseline
  2% gain in 8 weeks where BMI<20kg/m2; prevention of further weight loss where BMI>20kg/m2

SECONDARY OUTCOMES:
Muscle strength | Change over 8 weeks from baseline
  Hand grip strength
Food intake | Change over 8 weeks from baseline
  24-hour dietary recall
General appetite | Change over 8 weeks from baseline
  Likert scale assessment
Gastrointestinal tolerance | Change over 8 weeks from baseline
  Likert scale assessment
Serum electrolytes | Change over 4 weeks from baseline
Biscuit palatability | Change over 8 weeks from baseline
  Likert scale assessment
Compliance | Change over 8 weeks from baseline
  Self-reported diary

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Health and Social Care Trust, Londonderry, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No